CLINICAL TRIAL: NCT01518140
Title: Novel Oxygen Delivery Modalities for Refractory Dyspnea in Patients With Advanced Cancer
Brief Title: BiPAP-Vapotherm RCT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-0689
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Locally advanced; Recurrent; Metastatic disease; Oxygen Delivery Modalities; Shortness of breath; Dyspnea; VapoTherm; Bilevel positive airway pressure; BiPAP; Non-rebreather mask
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Dyspnea | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VapoTherm (Experimental): Participants receive air through VapoTherm for 1 hour, and then on an "as needed" basis for up to 4 hours. Participants then receive air through bilevel positive airway pressure (BiPAP) for up to 30 minutes, followed by 30 minutes using non-rebreather mask.
  Interventions: Device: Oxygen Delivery Devices; Behavioral: Questionnaires
- BiPAP (Experimental): Participants receive air through bilevel positive airway pressure (BiPAP) for 1 hour, and then on an "as needed" basis for up to 4 hours. Participants then receive air through VapoTherm for up to 30 minutes, followed by 30 minutes using non-rebreather mask.
  Interventions: Device: Oxygen Delivery Devices; Behavioral: Questionnaires
- Non-Rebreather Mask (Experimental): Participants receive air through Non-Rebreather Mask for 1 hour, and then on an "as needed" basis for up to 4 hours. Participants then receive air through VapoTherm for up to 30 minutes, followed by 30 minutes using bilevel positive airway pressure (BiPAP).
  Interventions: Device: Oxygen Delivery Devices; Behavioral: Questionnaires

INTERVENTIONS:
Device: Oxygen Delivery Devices — Participants receive air through VapoTherm for 1 hour, and then on an "as needed" basis for up to 4 hours. Participants then receive air through bilevel positive airway pressure (BiPAP) for up to 30 minutes, followed by 30 minutes using non-rebreather mask.
Behavioral: Questionnaires — 2 Questionnaires completed at baseline taking about 10 minutes to complete. At end of visit, questionnaire completion taking about 5 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if 3 breathing devices reduce feeling short of breath in cancer patients. Researchers also want to learn if these devices can help to control shortness of breath.

DETAILED DESCRIPTION:
Device A is designed to get more air in and out of their lungs without using as much effort as regular breathing. The air is given through a mask, and the amount of air can be set to different levels.

Device B is designed to deliver air in and out of the lungs. The air is warmed, filtered for bacteria, and then delivered through the nose using a tube under the nostrils.

Device C is designed to deliver air in and out of the lungs. The air is given through a mask, and the amount of air can be set to different levels.

Study Groups and Device Use:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 3 groups:

* If you are in Group 1, you will receive air through Device A for 1 hour, and then on an "as needed" basis for up to 4 hours. Then you will receive air through Device B for up to 30 minutes, followed by 30 minutes using Device C.
* If you are in Group 2, you will receive air through Device B for 1 hour, and then on an as needed basis for up to 4 hours. Then you will receive air through Device A for up to 30 minutes, followed by 30 minutes using Device C.
* If you are in Group 3, you will receive air through Device C for 1 hour, and then on an as needed basis for up to 4 hours. Then you will receive air through Device A for up to 30 minutes, followed by 30 minutes using Device B.

The study staff will help you use the devices. The maximum time allowed using the 3 devices is 6 hours total.

During the "as needed" use period (4 hours), you will switch between the device you were assigned to and the same air delivery device and oxygen level that you were using just before you started the study.

Study Visit:

During your study visit, the following tests and procedures will be performed:

* From your medical record, the study staff will collect information about your age, sex, race, disease type, how well you are able to perform the normal activities of daily living, any drugs you are taking, and possible causes of shortness of breath.
* You will complete 2 questionnaires. The first asks about breathing symptoms, and the second asks about other symptoms you may be having. It should take about 15 minutes to complete these questionnaires.
* Your heart rate, breathing rate, and blood pressure will be recorded.
* The level of air you breathe out will be recorded using a measuring device on your chest.
* Before and after using the devices, you will be asked how hard it is to catch your breath and about any side effects you may be having.
* At the end of the visit, you will fill out a questionnaire that asks about which device you prefer. It should take about 5 minutes to complete this questionnaire.

Length of Study:

You will be on this study for up to 6 hours. You will be taken off study and the device will be stopped if intolerable side effects occur while using a study device.

This is an investigational study. The 3 breathing devices are commercially available and FDA approved for delivering oxygen when medically needed, including in cancer patients. It is investigational to collect information from patients to rate how well the study devices may affect shortness of breath.

Up to 90 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced cancer, defined as locally advanced, recurrent, or metastatic disease
2. Persistent dyspnea, defined in this study as dyspnea at rest with an average intensity level >=3/10 on the numeric rating scale for at least 1 week and just prior to study initiation despite supplemental oxygen for at least 30 minutes
3. Dyspnea judged clinically to be predominantly due to the underlying malignancy, with or without obstructive lung disease
4. Inpatient at MD Anderson Cancer Center
5. Able to communicate in English
6. Expected life expectancy >1 week
7. Age 18 or older

Exclusion Criteria:

1. Hypoxia (i.e., O2 saturation <90%) despite supplemental oxygen at 15 L/min
2. Hemodynamic instability (systemic blood pressure (SBP) <90 mmHg) within 1 hour of study initiation
3. Comatose state or delirium, as indicated by a Memorial Delirium Assessment Scale score of 13 or higher
4. Uncontrolled arrhythmia as per clinical record at enrollment
5. Upper GI bleeding within 2 weeks of enrollment
6. Esophageal rupture at enrollment
7. Upper airway obstruction at enrollment
8. History of facial trauma within 2 weeks of enrollment
9. Facial, upper airway, or GI surgery within 2 weeks of enrollment
10. Thoracic surgery within 6 weeks of enrollment
11. Excessive airway secretions interfering with BiPAP administration
12. Undrained pneumothorax at enrollment
13. Partial or complete small bowel obstruction or severe nausea/vomiting (Edmonton symptom assessment scale nausea >7/10) within 48 hours of enrollment
14. Hemoglobin <8 g/dL at the time of enrollment (blood drawn within past 2 weeks)
15. Acute exacerbation of chronic obstructive pulmonary disease (COPD) or heart failure within 1 week of enrollment by history or physical
16. Known CO2 retainers as per clinic station
17. Known pulmonary hypertension as per clinic station
18. Unwillingness to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 3 Different Oxygen Delivery Methods | 6 hours
  Maximal inspiratory pressure measured at baseline, at end of the first hour, and after 4 hours of as-needed intervention using the NS 120-TRR negative inspiratory force monitor. Five consecutive efforts will be recorded, with a 1-minute pause between each effort (Ha-rik-Khan et al. 1998). Participants asked to rank the breathing devices based on their (1) efficacy in helping them to breathe, (2) comfort, and (3) ease of use on a numeric rating scale from 0 (best) to 10 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- [Derived] Hui D, Morgado M, Chisholm G, Withers L, Nguyen Q, Finch C, Frisbee-Hume S, Bruera E. High-flow oxygen and bilevel positive airway pressure for persistent dyspnea in patients with advanced cancer: a phase II randomized trial. J Pain Symptom Manage. 2013 Oct;46(4):463-73. doi: 10.1016/j.jpainsymman.2012.10.284. Epub 2013 Jun 2. PMID 23739633
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org